CLINICAL TRIAL: NCT04727281
Title: Dialysis Recovery Time: Associated Factors and Its Relation to Quality of Life in Hemodialysis Patients.
Brief Title: Dialysis Recovery Time: Associated Factors and Its Relation to Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, Assistant professor & lecturer, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Dialysis Recovery Time
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Dialysis; Complications
Keywords: dialysis, recovery time, fatigue, quality of life
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dialysis patients (Experimental): Patients included in the study will be recruited from the dialysis units in Alexandria University Hospitals.
  Interventions: Other: Quality of life assessment using the Kidney Disease Quality of Life 36 (KDQOL-36) short form and Malnutrition-Inflammation Score

INTERVENTIONS:
Other: Quality of life assessment using the Kidney Disease Quality of Life 36 (KDQOL-36) short form and Malnutrition-Inflammation Score — Data about nutritional status using the Malnutrition-Inflammation Score, and Quality of life assessment using the Kidney Disease Quality of Life 36 (KDQOL-36) short form. Dialysis related data, The time needed for the patient to recover from a dialysis session (in minutes), Detailed history taking, Thorough physical examination, Laboratory Investigations:
  • Hemoglobin , Serum sodium and potassium , Serum creatinine and blood urea , Serum phosphorus, serum calcium , Serum PTH level , Serum albumin ,CRP ,Total iron-binding capacity .

SUMMARY:
This study aims to identify factors affecting dialysis recovery time and the relation between dialysis recovery time and quality of life in hemodialysis patients.

DETAILED DESCRIPTION:
Dialysis is defined as the diffusion of molecules in solution across a semipermeable membrane along an electrochemical concentration gradient. The primary goal of hemodialysis (HD) is to restore the intracellular and extracellular fluid environment that is characteristic of normal kidney function. In addition to diffusion, solutes may pass through pores in the membrane by means of a convective process driven by hydrostatic or osmotic pressure gradients a process called ultrafiltration. During ultrafiltration, there is no change in solute concentrations; its primary purpose is the removal of excess total body water.

Fatigue is a well-known and frequent symptom in HD patients with a reported association with the decrease in health-related quality of life commonly found in this population. The prevalence of fatigue ranges from 60% to as high as 97% in patients on long-term renal replacement therapy. Despite this fact, health care providers are still unaware of both its presence and severity.

The clinical assessment of fatigue in dialysis patient can be somehow difficult for the treating physicians. Patients usually show diversity in their recovery from fatigue. However, early recognition is essential because a number of treatable causes can be easily identified.

Post-HD fatigue is a common incapacitating symptom affecting renal population. It is defined as a feeling of exhaustion that regularly follows each dialysis procedure. Uremia-related factors such as anemia, nutritional deficiency and enhanced inflammatory state could possibly lead to post-HD fatigue. In addition, the HD procedure itself including the efficiency of HD session, type of dialyzer and ultrafiltration rate are potential exacerbating factors for post-HD fatigue.

Several methods have been proposed as a way to assess post-HD fatigue with the "time to recover (minutes) from HD" being one of them. Lindsay et al. assisted patients' responses to the single open-ended question, "How long does it take you to recover from a dialysis session?".Lindsay et al. found that post hemodialysis recovery time is an important indicator for patients' quality of life.

Health-related quality of life (HRQOL) is a critically important outcome for patients with end-stage renal disease (ESRD). The National Quality Forum selected the Kidney Disease Quality of Life Short-Form survey (KDQOL™-36) as the tool of choice for assessing this outcome in adult patients with ESRD; assessment is required within 4 months of initiating dialysis, and annually thereafter. This 36-question survey instrument was published in 2000. The KDQOL™-36 contains 5 subscales: the Physical Component Summary(PCS), Mental Component Summary (MCS), Burden of Kidney Disease (BKD), Symptoms and Problems of Kidney Disease (SPKD), and Effects of Kidney Disease (EKD). The first 2 subscales are a general measure of HRQOL, whereas the last 3 assess issues specific to patients with ESRD or earlier stages of chronic kidney disease.(15) The Kidney Disease Quality of Life Short Form 36 (KDQOL-36) provides accurate estimate for fatigue severity and was previously used in HD population.

Although post-HD fatigue commonly exists in dialysis patients, it is usually underestimated by physicians. For this reason, appropriate and early identification of symptoms and associated factors might improve the patient's quality of life. Extending the research in this area will certainly be of great value to HD population.

ELIGIBILITY:
Inclusion Criteria:

* End Stage renal disease patients who have been assigned to regular long-term hemodialysis and perform thrice weekly, four hours HD sessions for more than 90 days.
* Patient's age of 18 years of more. They should be able to read and write, and in a complete mental health.

Exclusion Criteria:

* Inability to answer the questionnaires because of hearing or reading problems, dementia, actual instability of clinical conditions requiring hospitalization, liver failure, and active cancer.
* Patients who experience a decline in the level of consciousness during the HD session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
dialysis recovery time | 48-72 hours
  The time needed for the patient to recover from a dialysis session (in minutes).

SECONDARY OUTCOMES:
quality of life assessment | 90 days
  Quality of life assessment using the Kidney Disease Quality of Life 36 (KDQOL-36) short form.
nutritional status | 90 days
  Data about nutritional status using the Malnutrition-Inflammation Score

CONTACTS AND LOCATIONS:
Overall Officials: montasser M zeid, MD, Principal Investigator — Professor of Nephrology & Internal Medicine, Faculty of medicine, Alexandria University; mohamed mamdouh el sayed, MD, Study Chair — Lecturer of Nephrology & Internal Medicine, Faculty of medicine, Alexandria University; osama M Refai, MBBCh, Study Chair — resident of Nephrology & Internal Medicine, Alexandria University Hospitals
Locations (1):
- Faculty of Medicine, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Lindsay RM, Heidenheim PA, Nesrallah G, Garg AX, Suri R; Daily Hemodialysis Study Group London Health Sciences Centre. Minutes to recovery after a hemodialysis session: a simple health-related quality of life question that is reliable, valid, and sensitive to change. Clin J Am Soc Nephrol. 2006 Sep;1(5):952-9. doi: 10.2215/CJN.00040106. Epub 2006 Jul 6. PMID 17699312
- [Background] Sakkas GK, Karatzaferi C. Hemodialysis fatigue: just "simple" fatigue or a syndrome on its own right? Front Physiol. 2012 Jul 31;3:306. doi: 10.3389/fphys.2012.00306. eCollection 2012. No abstract available. PMID 22934057
- [Background] Rayner HC, Zepel L, Fuller DS, Morgenstern H, Karaboyas A, Culleton BF, Mapes DL, Lopes AA, Gillespie BW, Hasegawa T, Saran R, Tentori F, Hecking M, Pisoni RL, Robinson BM. Recovery time, quality of life, and mortality in hemodialysis patients: the Dialysis Outcomes and Practice Patterns Study (DOPPS). Am J Kidney Dis. 2014 Jul;64(1):86-94. doi: 10.1053/j.ajkd.2014.01.014. Epub 2014 Feb 14. PMID 24529994
- [Background] Cohen DE, Lee A, Sibbel S, Benner D, Brunelli SM, Tentori F. Use of the KDQOL-36 for assessment of health-related quality of life among dialysis patients in the United States. BMC Nephrol. 2019 Apr 1;20(1):112. doi: 10.1186/s12882-019-1295-0. PMID 30935377
- [Background] As'habi A, Tabibi H, Hedayati M, Mahdavi-Mazdeh M, Nozary-Heshmati B. Association of malnutrition-inflammation score, dialysis-malnutrition score and serum albumin with novel risk factors for cardiovascular diseases in hemodialysis patients. Ren Fail. 2015 Feb;37(1):113-6. doi: 10.3109/0886022X.2014.967615. Epub 2014 Oct 8. PMID 25296104
- [Derived] Elsayed MM, Zeid MM, Hamza OMR, Elkholy NM. Dialysis recovery time: associated factors and its association with quality of life of hemodialysis patients. BMC Nephrol. 2022 Sep 1;23(1):298. doi: 10.1186/s12882-022-02926-0. PMID 36050656